CLINICAL TRIAL: NCT00000982
Title: A Randomized Trial To Evaluate the Impact of Maintaining Steady-State Concentrations of Azidothymidine (AZT) Versus an Intermittent Schedule of AZT Delivery in Children With Symptomatic HIV Infection
Brief Title: A Study of Azidothymidine in HIV-Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 103; NCI 89 C-102C
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1996-10

CONDITIONS: Encephalopathies; HIV Infections
Keywords: Central Nervous System Diseases; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Brain Diseases; HIV Infections; Central Nervous System Diseases; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
AMENDED 07/07/93: To evaluate whether continuous infusion AZT will impact neurodevelopmental deficits associated with HIV infection or alter rate of encephalopathy progression in children who have failed to improve or shown progression of these deficits despite optimal AZT therapy.

AMENDED: To assess whether didanosine (ddI) will be better tolerated than AZT administered by either continuous intravenous delivery or oral administration (ddI arm removed per amended version).To determine whether ddI will achieve comparable clinical efficacy as the continuous intravenous route of delivery of AZT, and to assess whether either or both of these regimens are superior to that achieved with an intermittent AZT dosage schedule. To determine whether there are differences in patient or parent (guardian) compliance between the three treatment regimens. Original design: To determine whether the pharmacokinetic profile (bloodstream levels) of zidovudine (AZT) influences its effectiveness on HIV infection in children. That is, the study seeks to find out whether there is a difference in the effect of AZT when given as a continuous intravenous infusion (and, if available, an oral sustained release dose) compared to an intermittent (not continuous) dose given orally every 6 hours. The study also plans to determine (1) whether there are differences in the tolerance and side effects associated with AZT when given on an intermittent schedule as opposed to a steady-state schedule; (2) the extent of variation from patient to patient in AZT levels and whether the plasma and cerebrospinal fluid levels of AZT are related to the degree of therapeutic effectiveness; and (3) whether there are differences in the response of children who acquired HIV infection perinatally (just before, during, or just after the time of birth) versus those who acquired HIV infection by transfusion.

One of the most serious effects of HIV disease in children is neuropsychological deterioration (relating to mental and nervous system functioning). This complication affects the vast majority of HIV infected children. A previous study of continuous intravenous administration of AZT in pediatric patients with HIV infection showed consistent and dramatic improvements of symptoms in all patients that had shown neurodevelopmental deficits or abnormalities. These improvements were seen within 3 to 4 weeks after AZT treatment was started. Neurodevelopmental improvements have been sustained on AZT, usually showing steady improvement which, in some patients, was associated with restoration of pre-HIV intellectual and neurological function. This study also showed an increase in the IQ scores of children receiving continuous infusion of AZT who did not have overt clinical evidence of encephalopathy (disease of the brain). Thus changes in cognitive function may be among the earliest signs of AIDS encephalopathy and underscores the need to start therapies that will treat the central nervous system in patients who appear to be clinically intact. A study comparing continuous infusion to intermittent dosing of AZT showed a significant increase in IQ scores for those children receiving the continuous dose compared to those treated with the intermittent schedule. Although a portable infusion pump allows patients to receive continuous infusion of AZT, a sustained release oral formulation that could provide a continuous release of AZT into the bloodstream would be highly desirable.

DETAILED DESCRIPTION:
One of the most serious effects of HIV disease in children is neuropsychological deterioration (relating to mental and nervous system functioning). This complication affects the vast majority of HIV infected children. A previous study of continuous intravenous administration of AZT in pediatric patients with HIV infection showed consistent and dramatic improvements of symptoms in all patients that had shown neurodevelopmental deficits or abnormalities. These improvements were seen within 3 to 4 weeks after AZT treatment was started. Neurodevelopmental improvements have been sustained on AZT, usually showing steady improvement which, in some patients, was associated with restoration of pre-HIV intellectual and neurological function. This study also showed an increase in the IQ scores of children receiving continuous infusion of AZT who did not have overt clinical evidence of encephalopathy (disease of the brain). Thus changes in cognitive function may be among the earliest signs of AIDS encephalopathy and underscores the need to start therapies that will treat the central nervous system in patients who appear to be clinically intact. A study comparing continuous infusion to intermittent dosing of AZT showed a significant increase in IQ scores for those children receiving the continuous dose compared to those treated with the intermittent schedule. Although a portable infusion pump allows patients to receive continuous infusion of AZT, a sustained release oral formulation that could provide a continuous release of AZT into the bloodstream would be highly desirable.

AMENDED 07/07/93: Children with progressive encephalopathy who have received a minimum of 3 months of oral or intermittent AZT or who have failed to improve following 6 months of optimal AZT will receive continuous infusion AZT via a portable infusion pump.

AMENDED: The oral sustained release has been dropped and is now oral ddI. Added has been a planned stratification for randomization for patients who received any antiretroviral therapy 4 or more weeks prior to study entry. The informed consent was modified to reflect ddI toxicities from adult studies. Computerized Tomography radiation dosimetry is now included.

AMENDED: Dropping the ddI component and open only to children with encephalopathy meaning they are losing milestones, this is equal to a P2 CDC rating . Testing the difference in intermediate vs continuous AZT. 12/1990. Original design: Children are first evaluated for randomization according to whether they have or do not have evidence of neurodevelopmental deficits at the time of the initial pretreatment evaluation. Patients are assigned to 1 of 3 groups, to receive AZT (1) by continuous infusion; (2) by oral, intermittent (every 6 hours) dosing; or (3) by oral sustained-release dosing. If the oral sustained-release formulation is not available when this study begins, it will begin with only the first 2 groups. The sustained release preparation will be evaluated as soon as it is available. Patients will be tested to measure physical or biological improvement in neurodevelopmental function.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Steroids for children with lymphocytic interstitial pneumonitis (LIP) who are steroid dependent.
* Maintenance amphotericin B and antituberculosis chemotherapy.
* Immunoglobulin therapy for children who develop at least three serious bacterial infections while receiving zidovudine (AZT) therapy.
* Prophylactic therapy for children who have had a previous episode of Pneumocystis carinii pneumonia (PCP) and who are receiving such therapy.

AMENDED 07/07/93:

Only HIV-related encephalopathy patients eligible (i.e., children with progressive encephalopathy who have received a minimum of 3 months of oral or intermittent AZT or who have failed to improve following 6 months of optimal AZT).

ORIGINAL DESIGN:

Eligibility criteria used are similar to those being used in the "Multicenter Trial to Evaluate Oral Retrovir in the Treatment of Children with Symptomatic HIV Infection," currently Protocol 88 C-92a.

Children are included:

* With overt encephalopathy as well as those who may have a subclinical cognitive impairment.
* Children must have laboratory evidence of HIV infection as demonstrated by either a positive viral culture (blood or cerebrospinal fluid) or detectable serum P24 antigen or repeatedly positive test for HIV antibody. HIV antibody must be determined by federally licensed ELISA test and confirmed by Western blot.
* Children with AIDS or ARC must have at least one of the following laboratory criteria indicative of immunologic abnormality:
* Hypergammaglobulinemia (IgG or IgA) defined as immunoglobulin values greater than upper limit of the age-adjusted normal.
* Hypogammaglobulinemia (IgG or IgA) defined as immunoglobulin levels less than lower limit of the age-adjusted normal.
* Absolute depression in CD4+ cells of 500 cells/mm3 or less.
* Decreased helper/suppressor ratio of 1.0 or less.
* Depressed in vitro mitogen response to at least one antigen (pokeweed, phytohemagglutinin, concanavalin A, Staphylococcus aureus, tetanus toxoid, Candida).
* Parent or guardian available to give written informed consent.

Prior Medication:

Allowed within 4 weeks of study entry:

* Immunoglobulin for thrombocytopenia.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Serious bacterial, fungal, or parasitic infections requiring parenteral therapy, at the time of study entry.

Concurrent Medication:

Excluded:

* Clofazimine, ansamycin (or other experimental agents or agents that may modify zidovudine (AZT) toxicity or safety) for active chronic opportunistic infection at time of study entry.
* Chronic use of drugs that are metabolized by hepatic glucuronidation (and may alter the metabolism of AZT) (e.g., acetaminophen).
* Prophylaxis for Pneumocystis carinii pneumonia (PCP) for children who have not had a previous episode of PCP, oral candidiasis, or otitis media.
* Immunoglobulin therapy not specifically allowed.

Patients with the following are excluded:

* Serious bacterial, fungal, or parasitic infections requiring parenteral therapy, at the time of study entry.
* Lymphocytic interstitial pneumonitis (LIP) and no additional AIDS-defining indicator disease as specified in the CDC Surveillance Case Definition for AIDS.

Prior Medication:

Excluded within 4 weeks of study entry:

* Other antiretroviral agents including ribavirin, HPA-23, dideoxycytosine (ddC), soluble CD4, and dideoxyadenosine (ddA) / didanosine (ddI).
* Immunomodulating agents including steroids, interferon, isoprinosine, and IL-2 not specifically allowed.
* Immunoglobulin not specifically allowed.
* Excluded within 2 weeks of study entry:
* Any other experimental therapy.
* Drugs that cause prolonged neutropenia or significant nephrotoxicity.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Lymphocyte transfusion for immune reconstitution.
* Excluded within 3 months of study entry:
* Bone marrow transplant.

Risk Behavior:

Excluded:

* Active alcohol or drug abuse.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75
Dates: Primary Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pizzo PA, Study Chair
Locations (7):
- United States (7):
  - Children's Hosp of Washington DC / Children's Natl Med Ctr, Washington D.C., District of Columbia
  - Univ of Florida Med Ctr, Jacksonville, Florida
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Walter Reed / USUHS / Pediatrics, Bethesda, Maryland
  - Natl Cancer Institute / HIV / AIDS Malignancy Branch, Bethesda, Maryland
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - Duke Univ Med Ctr, Durham, North Carolina